CLINICAL TRIAL: NCT02053246
Title: Improving Treatment Personalization of Pulmonary Hypertension Associated With Diastolic Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study funding ended before recruitment completed.
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201501144 -N; K23GM112014 (NIH)
Record Dates: First submitted 2014-01-24; First posted 2014-02-03 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Hypertension; Diastolic Heart Failure; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure, Diastolic | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nebivolol (Experimental): Participants will be started at 2.5 mg of nebivolol by mouth daily if on a beta-blocker the dose will start at 5mg, and titrated up to 10 mg daily, as tolerated.
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Nebivolol will be started at 2.5 mg by mouth daily if on a beta-blocker the dose will start at 5mg, and titrated up to 10 mg daily, as tolerated.

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF), is one of the leading causes of pulmonary hypertension (PH). Despite the severity of this disease, no established treatments exist for this class of PH. Nebivolol is a drug used in high blood pressure and heart failure, but not used in patients with PH. Due to some additional properties it possesses, the investigators believe nebivolol will improve disease severity in patients with PH associated with HFpEF. The hypothesis of this research study is that nebivolol improves PH severity in patients with HFpEF, as measured by hemodynamic and clinical parameters.

DETAILED DESCRIPTION:
This research study will be a prospective, open-label 18-week clinical study of nebivolol in patients with PH associated with HFpEF. Patients will be identified in clinic based on echocardiogram (TTE) and right heart catheterization (RHC) results (both part of standard clinical care) indicating PH and HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years of age) with World Health Organization Group 2 Pulmonary Hypertension (Mean pulmonary artery pressure ≥ 25 mmHg and pulmonary capillary wedge pressure ≥ 15 mmHg)
* New York Heart Association class II-IV symptoms
* Left ventricular ejection fraction (LVEF) ≥ 45%

Exclusion Criteria:

* Other causes of heart failure other than diastolic dysfunction, such as restrictive cardiomyopathy or infiltrative cardiomyopathy
* Women who are pregnant or nursing
* Liver cirrhosis,
* Primary valvular disease
* Acute coronary syndrome
* Causes of PH other than that of heart failure, such as: chronic thromboembolic PH, sickle-cell disease, or sarcoidosis
* Severe bradycardia or greater than 1st degree heart block
* Decompensated heart failure
* Current use of a third generation beta-blocker (nebivolol, carvedilol, or labetalol) or high dose of any beta-blockers (greater than 100 mg daily of metoprolol, or equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Duarte, PharmD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol
Started | 11
Completed | 7
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nebivolol
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Weight [Mean (Standard Deviation); unit: kilograms] — Population: 2 patients withdrew before measurement
  kilograms
    number analyzed (Participants) | 9
    (all) | 93.0 (29.8)
Height [Mean (Standard Deviation); unit: cm] — Population: 2 patients withdrew before measurement
  cm
    number analyzed (Participants) | 9
    (all) | 164.6 (9.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 2 patients withdrew before measurement
  mmHg
    number analyzed (Participants) | 9
    (all) | 130.1 (16.0)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 2 patients withdrew before measurement
  mmHg
    number analyzed (Participants) | 9
    (all) | 68.0 (12.7)
Mean Pulmonary Artery Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 2 patients withdrew before measurement
  mmHg
    number analyzed (Participants) | 9
    (all) | 35.2 (7.2)
Pulmonary Artery Wedge Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 2 patients withdrew before measurement
  mmHg
    number analyzed (Participants) | 9
    (all) | 19.6 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Pulmonary Vascular Pressure
Description: Difference between baseline and 18 week mean pulmonary artery pressure and pulmonary artery wedge pressure
Time Frame: baseline - 18 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nebivolol
Number analyzed (Participants) | 7
mmHg
  Mean Pulmonary Artery Pressure Change | 0.43 (6.32)
  Pulmonary Artery Wedge Pressure Change | 1.0 (7.0)

2. Secondary Outcome: Changes in 6-minute Walk Distance
Description: Difference in 6-minute walk distance between baseline and 18 weeks.
Time Frame: baseline - 18 weeks
Population: Only patients who were able to complete walk tests at baseline and final study visits.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Nebivolol
Number analyzed (Participants) | 4
feet | -44.0 (299.8)

ADVERSE EVENTS:
Time Frame: Data were collected from enrollment until completion of final study visit at week 18.
Arm/Group | Nebivolol
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol (N=9)
Dizziness (General disorders) | 1 (1)
Fluid retention (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial was stopped prior to completion because funding ended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT02053246/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02053246/ICF_001.pdf